CLINICAL TRIAL: NCT03599375
Title: Safety and Clinical Activity of CD19 Chimeric Antigen Receptor T Cells in Treating Patients With Recurrent or Refractory CD19 Positive B Cell Acute Lymphoblastic Leukemia
Brief Title: Immunotherapy With CD19 CART-cells for B Cell Acute Lymphoblastic Leukemia
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: jiuwei cui (Other)
Responsible Party: Sponsor-Investigator, jiuwei cui, chief, The First Hospital of Jilin University
Organization: The First Hospital of Jilin University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FJLU-002
Record Dates: First submitted 2018-07-15; First posted 2018-07-26 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Leukemia, B-Cell
Keywords: Chimeric Antigen Receptor-Modified T Cells; CART; Recurrent B Cell Acute Lymphoblastic Leukemia; refractory B Cell Acute Lymphoblastic Leukemia; ALL
MeSH Terms: conditions — Leukemia, B-Cell; Burkitt Lymphoma

STUDY DESIGN:
Intervention Model Description: Patients with recurrent or refractory CD19+ ALL receive CD19 CAR T-cell immunotherapy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- B-ALL treated with CD19 CART cell (Experimental): The qualified CD19-targeted CART cells will be transferred to patient for 3 days as follow:D1,10% fraction;D2,30%;D3 60%. The number of CART cells for each course will be about 1×106/kg. If complete response (CR) or complete response with incomplete hemogram recovery (CRi) in hemogram is achieved after the first course of treatment, further treatment will be decided according to the clinical assessment and the wishes of the patient.If partial response (PR) is achieved after the first course, 1 or 2 courses of treatment will be continued. If there is no response (NR) after the first course, the treatment will be ceased or restarted based on the clinical assessment or patients' wishes. Treatent may be discontinued due to any severe toxicity, such as cytokine release syndrom.
  Interventions: Biological: CD19-targeted CART cells

INTERVENTIONS:
Biological: CD19-targeted CART cells — CD19 CAR T cells was transduced with a lentiviral vector to express anti-CD19 scFv.This is a second generation CRAT.

SUMMARY:
This study aims to evaluate the safety and clinical activity of CD19 Chimeric Antigen Receptor (CAR) redirected autologous T-cells in treating patients with recurrent or refractory CD19 positive B cell ccute lymphoblastic leukemia,and dynamically observe the changes of CAR-T in patients and the residual tumor.

DETAILED DESCRIPTION:
In this single-center, open-label, single-arm, prospective clinical trial, a total of 20 recurrent or refractory CD19+ B cell acute lymphoblastic leukemia patients will be enrolled.After recruiting eligible patients,autologous peripheral blood mononuclear cells(PBMCs) will be purified from whole blood.The CD3+ T cells were subsequently selected and re-stimulated by anti-CD3 and anti-CD28 monoclonal antibodies.T cells will be transduced with lentiviral vector for the generation of the CD19 CART cell and administered by i.v. injection.The purpose of current study is to determine the safety and clinical efficacy of CD19 CAR T cells therapy in patients with recurrent or refractory CD19+ ALL.

ELIGIBILITY:
Inclusion Criteria:

* Recurrent or refractory B cell derived acute lymphoblastic leukemia (ALL)
* Patients who have failed at least one line of a standard treatment without effective treatment measures at present
* CD19 expression on the surface of B-ALL cells must be detected
* KPS>80
* Life expectancy >3 months
* Patients must have adequate cardiac function (no electrocardiogram with obvious abnormality, LVEF≥50%),adequate pulmonary function as indicated by room air oxygen saturation of > 90%, and adequate renal function (Cr≤2.5 times of the normal range)
* The alanine aminotransferase (ALT) and the aspartate aminotransferase (AST)≤ 3 times of the normal range, and the total bilirubin (TBIL)≤2.0mg/dl(34.2umol/L)
* Hemoglobin(Hgb)≥80g/L
* Without contraindication of apheresis and cell isolation
* Patients and their families volunteer to participate in the research with signed written informed consent

Exclusion Criteria:

.Other concurrent severe and/or uncontrolled medical conditions: patients with another primary malignant disease; another severe and/or life-threatening medical disease.

* Evidence of uncontrolled current serious active infection
* HIV/HBV/HCV infection
* Pregnancy and nursing females
* Systemic glucocorticoid therapy within one week

Ages: 14 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-05-01 (Estimated); Primary Completion 2020-12-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
overall response rate(ORR) | Participants will be followed for the duration of the treatment, with an expected average of 3 months.
  ORR is defined as the proportion of partial responses plus complete responses.

SECONDARY OUTCOMES:
Progression free survival(PFS) | 15 years
  Progression-free survival is defined as the time from enrollment to first observation of progression or date of death (from any cause).
Overall survival(OS) | 15 years
  Overall survival, defined as the time from enrollment until death due to any cause. For patients who do not die, time to death will be censored at the time of last contact.